CLINICAL TRIAL: NCT03338244
Title: Mortality Reduction After Oral Azithromycin Contingency: Mortality Study
Acronym: MORDORIIMortY5
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: The Carter Center (Other); Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-01036-Y4; OPP1032340-A (Other Grant/Funding Number: The Bill and Melinda Gates Foundation)
Record Dates: First submitted 2017-11-07; First posted 2017-11-09 (Actual); Results first posted 2022-08-11 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-07

CONDITIONS: Childhood Mortality
Keywords: Childhood mortality; Mass treatment; Azithromycin; Infection
MeSH Terms: conditions — Infections | interventions — Azithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Azithro (Active Comparator): Communities will receive four rounds of biannual mass azithromycin.
  Interventions: Drug: Azithromycin
- Placebo (Placebo Comparator): Communities will receive four rounds of biannual mass placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Azithromycin — Children aged 1 month to 60 months per community will be offered weight or height-based, directly observed, oral azithromycin suspension every 6 months
  Other Names: Zithromax
  Arms: Azithro
Drug: Placebo — Children aged 1 month to 60 months per community will be offered weight or height-based, directly observed, oral placebo suspension every 6 months
  Arms: Placebo

SUMMARY:
MORDOR was a cluster-randomized placebo controlled trial that assessed the efficacy of mass azithromycin distributions for the prevention of childhood mortality. All communities were subsequently treated with mass azithromycin for one year. The present trial re-randomized communities to azithromycin or placebo for the fourth and fifth year of the study.

DETAILED DESCRIPTION:
Pre-trial treatments: in the original MORDOR trial, communities were randomized to 4 rounds of biannual mass distributions of either azithromycin or placebo (i.e, the first two years of the trial). All communities were subsequently treated with 2 rounds of biannual mass azithromycin (i.e., the fifth and sixth rounds, during the third year of the trial).

Present trial design: The present trial enrolls all communities previously enrolled in the Niger site of MORDOR, and re-randomizes communities to biannual mass distributions of either azithromycin or placebo (i.e., the seventh, eighth, ninth and tenth rounds of mass drug administration since randomization for the original MORDOR trial, occurring in the fourth and fifth year since randomization). This results in four patterns of community-based treatment: four years of azithromycin (AAAAA), three years of azithromycin followed by one year of placebo (AAAPP), two years of placebo followed by two years of azithromycin (PPAAA), and two years of placebo followed by one year of azithromycin and then one year of placebo (PPAPP). The primary outcome will be all-cause mortality in children aged 1-59 months,as determined by biannual census. The mortality rate following re-randomization (i.e., the seventh, eighth, ninth and tenth rounds of mass drug administration) will be compared between the two re-randomized groups.

ELIGIBILITY:
Inclusion Criteria:

* Communities- All communities eligible for MORDOR (NCT02047981)
* Individuals-All children aged 1-60 months (up to but not including the 5th birthday), as assessed via biannual census

Exclusion Criteria:

* Refusal of village chief (for village inclusion), or refusal of parent or guardian (for individual inclusion)

Ages: 1 Month to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66228 (Actual)
Dates: Start 2017-10-20 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tom M Lietman, MD, Principal Investigator — UCSF Proctor Foundation; Elodie Lebas, RN, Study Director — UCSF Proctor Foundation
Locations (2):
- UCSF Proctor Foundation, San Francisco, California, United States
- The Carter Center, Niamey, Niger

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: village
Period: Overall Study
Arm/Group | Azithro | Placebo
Started | 33173; 295 village | 33055; 297 village
Completed | 25995; 295 village | 25568; 297 village
Not Completed | 7178; 0 village | 7487; 0 village

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Azithro | Placebo | Total
Number analyzed (Participants) | 33173 | 33055 | 66228
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 33173 | 33055 | 66228
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16052 | 16084 | 32136
  Male | 17121 | 16971 | 34092
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 33173 | 33055 | 66228
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Niger | 33173 | 33055 | 66228

OUTCOME MEASURES:

1. Primary Outcome: All-cause Mortality Rate in Children Aged 1-60 Months
Description: as measured by presence on census and absence on sequential census due to death
Time Frame: 24 months
Population: Number of participants at the start of MORDOR III
Measure: Number (95% Confidence Interval); unit: deaths per 1000 person years
Arm/Group | Azithro | Placebo
Number analyzed (Participants) | 33173 | 33055
deaths per 1000 person years | 24.8 [23.1 to 26.5] | 26.7 [24.5 to 28.5]

2. Primary Outcome: Macrolide Resistance in Children Aged 1-60 Months
Description: as measured by nasopharyngeal swabs
Time Frame: 18 months
Population: We did collect nasopharyngeal swabs but pooling and DNA-seq that works with rectal samples was not sensitive enough for NP samples. So we have to wait for technology to catch up to be able to report these results.
Arm/Group | Azithro | Placebo
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Normalized Macrolide Resistance in Children Aged 1-60 Months
Description: as measured by rectal swabs. Fraction of macrolide resistance from stool specimens in children 1-60 months (core). For Niger, this includes RNA, DNA, and TAC-card methods (a binary outcome at the individual level).
Time Frame: 18 months
Population: 1,004 children in total (557 from 15 placebo-treated communities and 447 from 14 azithromycin-treated communities).
Measure: Mean (95% Confidence Interval); unit: reads per million (rM)
Arm/Group | Azithro | Placebo
Number analyzed (Participants) | 447 | 557
reads per million (rM) | 79.85 [44.31 to 124.14] | 15.79 [5.72 to 27.39]

4. Secondary Outcome: Microbial Composition of Stool
Description: as measured by Meta-genomic Deep Sequencing
Time Frame: 18 months
Population: Unfortunately, we didn't collect stool, so we won't be able to report this.
Arm/Group | Azithro | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Campylobacter and Other Pathogenic Organisms in Stool
Description: as measured by molecular techniques
Time Frame: 18 months
Population: Unfortunately, we didn't collect stool, so we won't be able to report this.
Arm/Group | Azithro | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 years
Description: No adverse events were reported other than death
Arm/Group | Azithro | Placebo
All-Cause Mortality (participants affected / at risk) | 1493/33173 | 1584/33055
Serious Adverse Events (participants affected / at risk) | 0/33173 | 0/33055
Other Adverse Events (participants affected / at risk) | 0/33173 | 0/33055

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-10-01): https://cdn.clinicaltrials.gov/large-docs/44/NCT03338244/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-01): https://cdn.clinicaltrials.gov/large-docs/44/NCT03338244/SAP_001.pdf